CLINICAL TRIAL: NCT03190057
Title: Evaluation of Effectiveness and Safety of BIOFREEDOM™ FAMILY Stent in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: IRIS-BioFreedom Cohort in the IRIS-DES Registry
Acronym: IRISBioFreedom
Status: Terminated | Type: Observational
Why Stopped: Funding issue
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Department of Medicine, Heart Institute, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2017-04
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Coronary Stenosis
Keywords: BioFreedom; Drug Eluting Stent; Coronary Artery Disease
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive percutaneous coronary intervention
  Interventions: Device: BIOFREEDOM™ FAMILY stent

INTERVENTIONS:
Device: BIOFREEDOM™ FAMILY stent — Percutaneous coronary intervention with BIOFREEDOM™ FAMILY stent

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of BIOFREEDOM™ FAMILY stent in the "real world" daily practice as compared with other drug-eluting stents.

DETAILED DESCRIPTION:
BIOFREEDOM™ FAMILY stent means that Biofreedom stent, Biofreedom Ultra and the other stents with names starting with Biofreedom.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Patient with BIOFREEDOM™ FAMILY stent
* Written consent

Exclusion Criteria:

* Intervention with BIOFREEDOM™ FAMILY stent and other drug eluting stent at the same time
* Life-expectancy less than 1 year
* Cardiac shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with BIOFREEDOM™ FAMILY stent
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Composite event rate of death, non-fatal myocardial infarction (MI), or Target- Vessel Revascularization (TVR) | 1 year

SECONDARY OUTCOMES:
All cause death | 5 year
Cardiac death | 5 year
Myocardial Infarction | 5 year
Composite event rate of death or myocardial infarction (MI) | 5 year
Composite event rate of cardiac death or myocardial infarction (MI) | 5 year
Target- Vessel Revascularization | 5 year
Target- Lesion Revascularization | 5 year
Stent thrombosis | 5 year
Stroke | 5 year
Procedural Success rate | 5 day
  defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization.

CONTACTS AND LOCATIONS:
Locations (8):
- South Korea (8):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soonchunhyang University Hospital, Cheonan, Cheonan
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hospital, Incheon
  - Inje University Pusan Paik Hospital, Pusan
  - Asan Medical Center, Seoul
  - Eulji General Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided